CLINICAL TRIAL: NCT04547998
Title: A Prospective Blinded Within-Subject Randomized Controlled Clinical Study to Investigate the Safety and Effectiveness of RECELL for Repigmentation of Stable Vitiligo Lesions
Brief Title: Clinical Study to Investigate the Safety and Effectiveness of RECELL for Repigmentation of Stable Vitiligo Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP009
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Phototherapy

STUDY DESIGN:
Masking Description: The Central Review Committee (CRC) will be blinded to treatment assignment when adjudicating data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All Participants (within patient control) (Experimental): Each participant will serve as their own Control, receiving both Control and Investigational Interventions randomly allocated to treatment of a portion of a depigmented vitiligo lesion.
  Interventions: Device: Control Intervention (UVB); Device: Investigational Interventions (Ablative Laser Resurfacing + RECELL + UVB)

INTERVENTIONS:
Device: Control Intervention (UVB) — Targeted narrowband-UVB phototherapy in alignment with published Vitiligo Working Group recommendations.
  Other Names: Phototherapy
Device: Investigational Interventions (Ablative Laser Resurfacing + RECELL + UVB) — Spray-On Skin™ Cells prepared using RECELL will be applied to an area prepared by ablative laser, followed by targeted narrowband UVB phototherapy.

SUMMARY:
This is a prospective blinded within-subject randomized study to evaluate the application of Spray-On Skin™ Cells, prepared using the RECELL® Device for safe and effective repigmentation of ablated stable vitiligo lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Focal, segmental or generalized (i.e., nonsegmental) stable vitiligo, defined as no new depigmented areas nor any depigmented areas that have expanded in size within the preceding 12 months, regardless of whether the areas are intended to be used as study areas.

1a. Photo documentation (current and at least 12 months prior) of the patient's depigmented areas have been evaluated as stable by an independent Screening Committee.

2. The patient has not undergone topical treatment (e.g., steroids, tacrolimus) for the study areas within the past 90 days.

3. The patient has not undergone phototherapy (e.g., NB-UVB) for the study areas within the past 90 days.

4. The patient is a candidate for surgical intervention of a depigmented area, defined as a patient who has previously been compliant with but has not satisfactorily responded to both

a. topical therapy and b. a minimum of 3 months of phototherapy.

5. The patient must have two study areas available for treatment that:

1. are of similar size (±50%),
2. are between 16cm2 and 456cm2 (contiguous),
3. are similarly sun exposed,
4. have the same extent of leukotrichia, and
5. are judged clinically as ≥90% depigmented (by area).

   6. The patient is 18 years of age or older.

   7. The patient is willing and able to comply with post-treatment at-home phototherapy and all follow-up evaluations required by the study protocol.

   8. The patient agrees to abstain from any other treatment of the study areas for the duration of his/her participation in the study (52 weeks).

   9. The patient agrees to abstain from enrollment in any other interventional clinical trial for the duration of his/her participation in the study (52 weeks).

   10. In the opinion of the investigator, the patient must be able to:

a. Understand the full nature and purpose of the study, including possible risks and adverse events, b. Understand instructions, and c. Provide voluntary written informed consent.

Exclusion Criteria:

1. The study areas selected have concomitant dermatologic conditions other than vitiligo.
2. The study area selected for treatment includes the lips, eyelids, plantar surface of feet, palmar surface of hands, fingertips, wrists, ankles, elbows, or knees.
3. The patient is unable to undergo the treatment area preparation.
4. Patients who are pregnant.
5. Patients with:

   1. universalis vitiligo,
   2. depigmented areas over >30% of their body surface area,
   3. depigmented lips and fingertips (lip-tip vitiligo), or
   4. > 3 depigmented fingertips, defined as depigmentation of the dorsal aspect of the fingertip from the distal interphalangeal joint to the tip of the digit.
6. Patients with recent history (within previous 12 months) of:

   1. Koebnerization,
   2. confetti-like, or
   3. trichrome lesions.
7. Patients with a history of keloid formation.
8. Patients who have used a tanning salon in the past 60 days.
9. The patient has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives.
10. Current use of medications (e.g., anticoagulants such as heparin or warfarin) that in the investigator's opinion may compromise patient safety or trial objectives.
11. The patient has a known hypersensitivity to trypsin or compound sodium lactate for irrigation (Hartmann's) solution.
12. Life expectancy is less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of California, Irvine, Irvine, California
  - University of California, Davis, Sacramento, California
  - West Dermatology, San Diego, California
  - DMR Research, Westport, Connecticut
  - Skin Care Research, LLC, Hollywood, Florida
  - Miami Dermatology and Laser Institute, Miami, Florida
  - University of Massachusetts, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas at Austin Dell Medical School, Austin, Texas
  - Heights Dermatology, Houston, Texas

REFERENCES:
- [Background] Liu JP, Hsueh HM, Hsieh E, Chen JJ. Tests for equivalence or non-inferiority for paired binary data. Stat Med. 2002 Jan 30;21(2):231-45. doi: 10.1002/sim.1012. PMID 11782062

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The design of this study is a within-patient comparison. Protocol enrollment is 25 (participants), with 50 interventions (2 per patient).
Units Other Than Participants: depigmented vitiligo lesions
Groups:
- Control Intervention (UVB): A portion of each participant's vitiligo lesion is randomly assigned to receive the Control Intervention (within-patient control): Targeted narrowband-UVB (only)
- Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB): A portion of each participant's vitiligo lesion is randomly allocated to receive the Investigational Treatment: Spray-On Skin™ Cells prepared using RECELL will be applied to an area prepared by ablative laser, followed by targeted narrowband UVB phototherapy.
Period: Overall Study
Arm/Group | Control Intervention (UVB) | Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB)
Started | 25; 25 depigmented vitiligo lesions | 25; 25 depigmented vitiligo lesions
Completed | 25; 25 depigmented vitiligo lesions | 25; 25 depigmented vitiligo lesions
Not Completed | 0; 0 depigmented vitiligo lesions | 0; 0 depigmented vitiligo lesions

BASELINE CHARACTERISTICS:
Population: Experimental: All Participants (within patient control)
Groups:
- All Participants (Within Patient Control): All subjects will receive both RECELL and NV-UVB. Each subject will serve as their own Control, with a depigmented area receiving no RECELL treatment but receiving the same targeted NB-UVB as the investigational treatment area. Study treatment areas will be randomly assigned as Area A and Area B. Investigational treatment (RECELL) will be randomly allocated to either Area A or Area B.
  Spray-On Skin™ Cells 1:20 followed by NB-UVB: Skin cell suspension at expansion ratio 1:20 (donor area : recipient area), prepared using the RECELL System, will be applied to an ablated (de-epithelialized) area of depigmentation, followed by targeted phototherapy using NB-UVB.
  NB-UVB only: Each subject will serve as their own control, with a portion (or similar) depigmented lesion receiving the same targeted NB-UVB without application of skin cell suspension.
Arm/Group | All Participants (Within Patient Control)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of ≥80% Study Area Repigmentation
Description: Repigmentation was evaluated by qualified members of a Central Review Committee.
Time Frame: Week 24
Population: ITT
Measure: Number; unit: study areas
Units Other Than Participants: depigmented vitiligo lesions
Groups:
- Control Intervention (UVB): A portion of each participant's vitiligo lesion is randomly assigned to receive the Control Intervention (within-patient control): Targeted narrowband-UVB phototherapy (only)
Arm/Group | Control Intervention (UVB) | Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB)
Number analyzed (Participants) | 25 | 25
Number analyzed (depigmented vitiligo lesions) | 25 | 25
study areas | 0 | 9
Statistical Analysis 1: Comparison: Control Intervention (UVB) vs Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB); Test type: Superiority — The difference in the proportion of responders (RECELL-Control) was tested for superiority of RECELL treatment (with a 10% superiority margin). For the null hypothesis to be rejected and super-superiority of RECELL to Control to be established, the lower limit of the 2-sided 95% CI of the difference in the proportion of responders (RECELL-Control) had to be greater than 10%; p = 0.012, continuity-corrected method; Liu et al 2002

2. Secondary Outcome: Repigmentation Category
Description: Expert Central Review Committee categorization of the amount of area repigmented (0-25%, 26-50%, 51-79% and 80-100%). This is visual estimation of the vitiligo lesion area that has repigmented, with reference to training images. Higher %repigmentation is a better outcome.
Time Frame: Week 24
Population: ITT
Measure: Number; unit: depigmented vitiligo lesions
Units Other Than Participants: depigmented vitiligo lesions
Arm/Group | Control Intervention (UVB) | Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB)
Number analyzed (Participants) | 25 | 25
Number analyzed (depigmented vitiligo lesions) | 25 | 25
depigmented vitiligo lesions
  Repigmentation Category: 0% | 5 | 3
  Repigmentation Category: 1 to 25% | 13 | 6
  Repigmentation Category: 26 to 50% | 4 | 2
  Repigmentation Category: 51 to 79% | 3 | 5
  Repigmentation Category: 80 to 99% | 0 | 9
  Repigmentation Category: 100% | 0 | 0
Statistical Analysis 1: Comparison: Control Intervention (UVB) vs Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — P-value based on Wilcoxon signed rank test at 2-sided 0.05 significance level. The Wilcoxon signed rank test was based on the following repigmentation categories: 0% to 25%, 26% to 50%, 51% to 79%, and 80% to 100%

3. Secondary Outcome: Color Matching
Description: The Expert Central Review Committee visually judged the quality of repigmentation in terms of how closely it matches with the normal pigmentation seen in the surrounding area. The rating scale consists of poor, moderate, good, and excellent. Color matching can only be evaluated in instances of >0% repigmentation.
Time Frame: Week 24
Population: ITT
Measure: Number; unit: study areas with >0% repigmentation
Units Other Than Participants: study areas with >0% repigmentation
Groups:
- Control Intervention(UVB): A portion of each participant's vitiligo lesion is randomly assigned to receive the Control Intervention (within-patient control): Targeted narrowband-UVB phototherapy (only)
Arm/Group | Control Intervention(UVB) | Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB)
Number analyzed (Participants) | 25 | 25
Number analyzed (study areas with >0% repigmentation) | 20 | 22
study areas with >0% repigmentation
  Color Matching Category: Poor | 0 | 1
  Color Matching Category: Moderate | 4 | 6
  Color Matching Category: Good | 12 | 9
  Color Matching Category: Excellent | 4 | 6
Statistical Analysis 1: Comparison: Control Intervention(UVB) vs Investigational Intervention (Ablative Laser Resurfacing + RECELL + UVB); Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney) — 2-sided (0.05 significance level), based on 19 participants with assessable color matching outcomes for both treatments

ADVERSE EVENTS:
Time Frame: 52 Weeks
Groups:
- Control Intervention: All subjects will receive both RECELL and NV-UVB. Each subject will serve as their own Control, with a depigmented area receiving no RECELL treatment but receiving the same targeted NB-UVB as the investigational treatment area. Study treatment areas will be randomly assigned as Area A and Area B. Investigational treatment (RECELL) will be randomly allocated to either Area A or Area B.
  Control area intervention: NB-UVB only without application of skin cell suspension.
- Investigational Intervention (RECELL): All subjects will receive both RECELL and NV-UVB. Each subject will serve as their own Control, with a depigmented area receiving no RECELL treatment but receiving the same targeted NB-UVB as the investigational treatment area. Study treatment areas will be randomly assigned as Area A and Area B. Investigational treatment (RECELL) will be randomly allocated to either Area A or Area B.
  Investigational Intervention: Spray-On Skin™ Cells 1:20 followed by NB-UVB: Skin cell suspension at expansion ratio 1:20 (donor area : recipient area), prepared using the RECELL System, will be applied to an ablated (de-epithelialized) area of depigmentation, followed by targeted phototherapy using NB-UVB.
Arm/Group | Control Intervention | Investigational Intervention (RECELL)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 5/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Intervention (N=25) | Investigational Intervention (RECELL) (N=25)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT04547998/Prot_SAP_002.pdf